CLINICAL TRIAL: NCT06674135
Title: Evaluating the Impact of Introducing Basaglar, a Long-acting Analog Insulin, on Clinical and Quality of Life Outcomes in Youth with Diabetes in Bangladesh
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Life for a Child Program, Diabetes Australia (Other)
Collaborators: Bangladesh Institute of Research and Rehabilitation in Diabetes, Endocrine and Metabolic Disorders (Other); BADAS-Centre for Health Research and Implementation (Unknown); Diabetic Association of Bangladesh (BADAS) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BADAS-ERC/EC/22/00325
Record Dates: First submitted 2024-11-03; First posted 2024-11-05 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Type I Diabetes
Keywords: Analog insulin; Basaglar; Bangladesh; Children and Adolescents; Type 1 diabetes; insulin pen-devices
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Introduction of Basaglar to insulin treatment regimen (Experimental): Switched to once daily injection of biosimilar insulin glargine via reusable pen and three mealtime bolus insulin injections of short-acting human insulin via needle and syringe
  Interventions: Drug: biosimilar insulin glargine

INTERVENTIONS:
Drug: biosimilar insulin glargine — Switched to once daily injection of biosimilar insulin glargine via reusable pen and three mealtime bolus insulin injections of short-acting human insulin via needle and syringe
  Other Names: Basaglar

SUMMARY:
This study aimed to determine the effect of introducing Basaglar and insulin pen injection devices on clinical and quality of life (QOL) parameters in children and young adults with type 1 diabetes in Bangladesh

DETAILED DESCRIPTION:
Analog insulins are widely used in middle- and high-income countries. However, use of analog insulin remains limited in lower-income countries due to their increased cost and lack of access, and human insulin remains the mainstay of treatment in these settings.

Long-acting (basal) analog insulin such as glargine have the benefit of a longer duration (up to 24 hours) and a minimal peak action, and generally, only one injection per day is required. Although glargine insulin has been shown to reduce the risk of overnight hypoglycemia, consistent improvement in blood glucose control (measured by HbA1c) when compared to human insulin has not been shown, and its impact on quality of life is also inconclusive. Furthermore, these studies have all been done in highly resourced countries.

Life for a Child (LFAC) provides diabetes supplies (insulin, syringes, meters and strips for blood glucose self-monitoring), diabetes-related education, mentoring and technical support to the team managing youth with type 1 diabetes (T1D) managed at the Bangladesh Institute of Research and Rehabilitation in Diabetes, Endocrine and Metabolic Disorders (BIRDEM) Hospital in Dhaka, Bangladesh. In 2022, LFAC commenced supplying Basaglar (glargine) insulin with insulin pen devices (HumaPen Ergo ll). This provided a unique opportunity to investigate the effect of introducing glargine (Basaglar) insulin in the low-resource setting of Bangladesh.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 1 diabetes (T1D). Diabetes was diagnosed in accordance with World Health Organization (WHO) criteria. Determination of diabetes type was made by the local investigators according to available clinical features and history: T1D was diagnosed upon abrupt onset of typical symptoms of diabetes with insulin required from diagnosis, and no acanthosis nigricans. They were usually non-obese.
* Duration of T1D at enrolment >12 months
* Aged 10-25 years (inclusive) at time of enrolment
* Current insulin regimen consisting of Humulin NPH® and R, or pre-mixed insulin (30/70 R/NPH), with no prior use of analogue insulin
* Attending Life for a Child, BIRDEM Hospital, Dhaka for their usual diabetes care

Exclusion Criteria:

• Previous use of analog insulin

Ages: 10 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 202 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Mean and median HbA1c (% and mmol/mol) | Baseline, 3-, 6-, 9- and 12-month follow-up visits
  HbA1c was measured at each study time point using the Minicap Sebia Autoanalyzer with venous blood

SECONDARY OUTCOMES:
Proportion of participants experiencing episodes of diabetic ketoacidosis | Baseline, 3-, 6-, 9- and 12-month follow-up visits
  Diabetic ketoacidosis was defined as hyperglycaemia (BGL>11mmol/L/200mg/dL) with a venous pH<7·3 or serum bicarbonate <15mmol/L and ketonaemia and ketonuria
Proportion of participants experiencing episodes of severe hypoglycaemia | Baseline, 3-, 6-, 9- and 12-month follow-up visits
  Severe hypoglycaemia was defined as an event with severe cognitive impairment (with or without coma and convulsions) requiring assistance by another person to administer carbohydrates, glucagon, or intravenous dextrose to restore glycaemia
Diabetes Quality of Life for Youth scale - Short Form (DQOLY-SF) | Baseline, 6- and 12-month follow-up visits
  The 21- item Diabetes Quality of Life in Youth - Short Form scale [1] was administered to participants to assess their health-related quality of life after the change in their insulin treatment regimen.
  Each item has 5 possible scores with a value from 0 to 4, with 0 representing "never" and 4 "all the time". Higher scores represent a higher impact of diabetes and a poorer quality of life; lower scores indicate greater quality of life. The highest possible score is 84 (21 x 4 i.e. "all the time" for all 21 items) and lowest possible score is 0 (21 x 0 i.e. "never" for all 21 items)
Participant self-reported satisfaction | 12-month follow-up visit
  A 5-item structured questionnaire was administered to participants in the intervention group to evaluate their satisfaction with the new insulin regimen, experience of using reusable insulin pens, and their experience of hypo- and hyperglycaemic episodes over the study period

CONTACTS AND LOCATIONS:
Overall Officials: Dr Bedowra Zabeen, MBBS, FCPS(Paediatrics), FRSPH, Principal Investigator — Life For a Child Program, BIRDEM, BADAS, Bangladesh
Locations (1):
- BIRDEM, the Bangladesh Institute of Research and Rehabilitation in Diabetes, Endocrine and Metabolic Disorders, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No
Due local privacy regulations, individual de-identified participant data will not be shared

REFERENCES:
- [Background] Skinner TC, Hoey H, McGee HM, Skovlund SE; Hvidore Study Group on Childhood Diabetes. A short form of the Diabetes Quality of Life for Youth questionnaire: exploratory and confirmatory analysis in a sample of 2,077 young people with type 1 diabetes mellitus. Diabetologia. 2006 Apr;49(4):621-8. doi: 10.1007/s00125-005-0124-0. Epub 2006 Jan 26. PMID 16525844